CLINICAL TRIAL: NCT04226950
Title: A Prospective, Single-center Clinical Trial of Pegylated Interferon Alfa-2b Versus Interferon Alfa Therapy in the Treatment of Childhood and Adolescent Essential Thrombocythemia
Brief Title: Pegylated Interferon Alfa-2b Versus Interferon Alfa Therapy in Childhood and Adolescent Essential Thrombocythemia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT2019001
Record Dates: First submitted 2019-12-10; First posted 2020-01-13 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-04

CONDITIONS: Essential Thrombocytopenia
Keywords: Essential Thrombocythemia; Childhood; Interferon Alfa; Pegylated Interferon Alfa-2b; Adolescent
MeSH Terms: conditions — Thrombocythemia, Essential | interventions — peginterferon alfa-2b

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant Interferon Alpha (Active Comparator): Recombinant Interferon Alpha, with an initial dose of 300 wu twice a week. Other interferons that have been listed can be used if Recombinant Interferon Alpha (300 wu) is not available, and the specific dose will be determined by the researchers.
  Interventions: Drug: Recombinant Interferon Alpha
- Pegylated Interferon Alfa-2b (Experimental): Pegylated Interferon Alfa-2b, with an initial dose of 135 ug once a week (body surface area < 1.73 m2) or 180 ug once a week ( body surface area≥1.73 m2).
  Interventions: Drug: Pegylated interferon alfa-2b

INTERVENTIONS:
Drug: Recombinant Interferon Alpha — Recombinant Interferon Alpha, with an initial dose of 300 wu twice a week. Other interferons that have been listed can be used if Recombinant Interferon Alpha (300 wu) is not available, and the specific dose will be determined by the researchers;
  Arms: Recombinant Interferon Alpha
Drug: Pegylated interferon alfa-2b — Pegylated Interferon Alfa-2b, with an initial dose of 135 ug once a week (body surface area < 1.73 m2) or 180 ug once a week ( body surface area≥1.73 m2).
  Arms: Pegylated Interferon Alfa-2b

SUMMARY:
Objectives: To compare the efficacy and safety in childhood and adolescent patients (<20 years) diagnosed as essential thrombocythemia treated with the Pegylated Interferon Alfa-2b vs. Interferon Alfa.

Study Design: A prospective, open-label, nonrandomized, single-center clinical trial

DETAILED DESCRIPTION:
This is a prospective, open-label, nonrandomized, single-center clinical trial between Interferon Alfa and Pegylated Interferon Alfa-2b in childhood and adolescent essential thrombocythemia (<20 years).

Patients will be divided into the following two treatment groups: 1. Recombinant Interferon Alpha, with an initial dose of 300 wu twice a week. Other interferons that have been listed can be used if Recombinant Interferon Alpha (300 wu) is not available, and the specific dose will be determined by the researchers; 2. Pegylated Interferon Alfa-2b, with an initial dose of 135 ug once a week (body surface area < 1.73 m2) or 180 ug once a week ( body surface area≥1.73 m2).

The current drug therapies and possible risks of Pegylated Interferon Alfa-2b and Interferon Alfa in the treatment of childhood and adolescent essential thrombocythemia will be fully introduced to the guardians (childhood patients) or patients (adolescent patients) by the researchers. Then the patients will be divided into one of the two groups according to the guardians' (childhood patients) or patients' (adolescent patients) will.

The dosage will be adjusted according to the results of laboratory examinations and patient tolerance. The patient will be transferred to the other group if intolerance or resistance occurs.

ELIGIBILITY:
Inclusion Criteria:

* <20 years old
* Male or Female
* Diagnosis of essential thrombocythemia according to the 2016 WHO criteria.
* Platelet count ≥ 450 × 109 / L for more than 6 months（If the patient has JAK2 V617F, CALR or MPL gene mutation, the history may be less than 6 months）
* Platelet count ≥ 1000 × 109 / L or other therapeutic indications at screening.
* The guardians has provided written informed consent prior to enrollment

Exclusion Criteria:

* Known to meet the criteria for primary myelofibrosis or polycythemia vera by 2016 WHO criteria
* Presence of any life-threatening co-morbidity
* Secondary thrombocytosis
* Familial thrombocytosis
* Resistance, or intolerance, or any contraindications to interferon
* Interferon is used in the past 1 month before enrollment
* Patients with previous or present thrombosis or active bleeding
* WBC<4× 109 / L
* HGB<110g/L
* Poor control of thyroid dysfunction
* Patients with a prior malignancy within the last 3 years
* Patients with severe cardiac or pulmonary dysfunction
* Severe renal damage (creatinine clearance < 30 ml / min)
* Severe liver dysfunction (ALT or AST > 2.5×ULN)
* Patients diagnosed as diabetes with poor control
* Patients with hepatitis B virus, hepatitis C virus replication or HIV infection
* Patients with a history of drug / alcohol abuse (within 2 years before the study)
* Patients that have participated in other experimental researches within one month before enrollment
* History of psychiatric disorder
* Any other circumstances that the investigator considers that the patient is not suitable to participate in the trial

Max Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-01-10 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-11-20 (Estimated)

PRIMARY OUTCOMES:
Change in platelet count | From the start of study treatment (Day 1) up to the end of month 12
  Proportion of subjects with a continuous platelet count ≤600×109/L or decrease ≥50% (<1000×109/L ) (at least 12 weeks) from baseline during treatment will be evaluated.

SECONDARY OUTCOMES:
The complete hematologic response rates | From the start of study treatment (Day 1) up to the end of month 12
  To compare the complete hematologic response rates between different treatment groups
Time to response in platelet count | From the start of study treatment (Day 1) up to the end of month 12
  Time to response in platelet count (<600×109/L) between different treatment groups
Impact of therapy on key biomarkers | From the start of study treatment (Day 1) up to the end of month 12
  To compare the proportion of subjects that display change on key biomarkers of the disease- JAK2V617F, CALR, MPL mutations.
Incidence of major cardiovascular and thrombotic events | From the start of study treatment (Day 1) up to the end of month 12
  To estimate incidence of major cardiovascular and thrombotic events (defined as cardiovascular death, myocardial infarction, stroke, transient ischemic attack, pulmonary embolism, Budd Chiari syndrome, deep vein thrombosis, and any other clinically relevant thrombotic event) while on active treatment or observation following end of treatment between different treatment groups
Incidence of development of myelodysplastic disorders, myelofibrosis, or leukemic transformation. | From the start of study treatment (Day 1) up to the end of month 12
  To estimate incidence of development of myelodysplastic disorders, myelofibrosis, or leukemic transformation between different treatment groups
Change in Myeloproliferative Neoplasm Symptom Assessment Form total symptom score | 12 months
  To compare the proportion of subjects that display change in Myeloproliferative Neoplasm Symptom Assessment Form total symptom score (0-100 scores, higher scores mean a worse outcome) between different treatment groups.
Specific pre-defined toxicity | From the start of study treatment (Day 1) up to the end of month 12
  To compare incidence of specific pre-defined toxicity including fatigue, flu-like symptoms, dizziness, injection site necrosis, dyspnea, pain, depression, blurred Vision, insomnia, anorexia, weight Loss, weakness, pruritis, sweating, fever, decreased Libido, hot Flashes, flushing.
Impact of therapy on bone marrow histopathology (selectable) | From the start of study treatment (Day 1) up to the end of month 12
  To compare the proportion of subjects that display change on bone marrow histopathology
Impact of therapy on cytogenetic abnormalities (selectable) | From the start of study treatment (Day 1) up to the end of month 12
  To compare the proportion of subjects that display change on cytogenetic abnormalities.
Death while on active treatment or observation following end of treatment | From the start of study treatment (Day 1) up to the end of month 12
  To compare the incidence of death while on active treatment or observation following end of treatment
Change in platelet count | From the start of study treatment (Day 1) up to the end of month 12
  Proportion of subjects with a continuous platelet count <1000×109/L in those with platelet count ≥1000×109/L before treatment (at least 12 weeks) will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Lei Zhang, MD, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China; Rongfeng Fu, Principal Investigator — Institute of Hematology & Blood Diseases Hospital, China
Locations (1):
- Institute of Hematology & Blood Diseases Hospital, Tianjin, Tianjin Municipality, China